CLINICAL TRIAL: NCT05672992
Title: Spatial Frequency Domain Imaging, Comparison of a Novel Method to Quantify Skin Fibrosis With Currently Used Methods in Scleroderma
Brief Title: Longitudinal Spatial Frequency Domain Imaging Study
Acronym: SFDI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Scleroderma Clinical Trials Consortium (SCTC) (Unknown); Fibrosis ARC: Connecting Tissues and Investigators (FCTI ARC) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-43177
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Systemic Scleroderma
Keywords: Spatial frequency domain imaging (SFDI); modified Rodnan skin score (mRSS); Skin biopsy; Skin fibrosis; Scleroderma skin patient reported outcome (SSPRO); Durometry; Ultrasound
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scleroderma Participants (Experimental): Participants in this arm will be asked to complete the Fitzpatrick skin type questionnaire to quantify skin tone and will have measurements taken with a colorimeter on the right and left forearms, hands, and fingers to quantify skin tone at the first study visit. Participants will be asked to complete the SSPRO questionnaire at the time of enrollment and every three months for the first 12 months and then every six months until the end of the study. At each study visit, a physician will measure the mRSS, which is a method of quantifying skin fibrosis; SFDI measurements, ultrasound, and durometry will then be done. Skin biopsies will be collected from the forearm of each subject annually. A small amount of blood will also be collected from subjects once per year to explore serum biomarkers of fibrosis.
  Interventions: Other: Spatial-frequency domain imaging (SFDI)
- Healthy controls (Active Comparator): Participants in this arm will be asked to complete the Fitzpatrick skin type questionnaire to quantify skin tone and will have measurements taken with a colorimeter on the right and left forearms, hands, and fingers to quantify skin tone at the first study visit. At each study visit, SFDI measurements, ultrasound, and durometry will be done. Skin biopsies will be collected from the forearm of each subject annually. A small amount of blood will also be collected from subjects once per year to explore serum biomarkers of fibrosis.
  Interventions: Other: Spatial-frequency domain imaging (SFDI)

INTERVENTIONS:
Other: Spatial-frequency domain imaging (SFDI) — SFDI is a method using near-infrared (NIR) light to generate wide field images (>10 x 10 cm) of tissue optical properties (absorption and scattering coefficients) at sub-surface depths of 1-10 mm. With SFDI the tissue surface (skin) is illuminated by a rapid sequence of sinusoidal light patterns of varying spatial frequency and at different optical wavelengths. Collected camera images are then processed to yield maps of sub-surface optical properties.

SUMMARY:
Scleroderma (SSc) is an autoimmune disease characterized by fibrosis (or collagen deposition) of the skin and internal organs. The extent of skin fibrosis is an important predictor of internal organ complications and increased mortality. Currently imprecise and subjective methods that varies amongst different doctors for the same patient are available to quantify skin fibrosis in patients, by "pinching" their skin and assessing how thick it is; this is the method used to determine the modified Rodnan skin score (mRSS).

Skin thickness and the amount of fibrosis can change over time due to disease progression or in response to therapy. In this research, longitudinal measurements will be taken to determine if spatial frequency domain imaging (SFDI) can detect changes in skin thickness that occur over time in response to therapy or from disease progression in scleroderma patients.

This study will compare SFDI with other clinical outcome assessments of skin thickness and fibrosis in scleroderma patients including mRSS, skin biopsy histology, scleroderma skin patient reported outcome (SSPRO), ultrasound, and durometry (durometer measures skin hardness). SFDI information will also be compared with capillaroscopy (allows for non-invasive imaging of the nailfold capillaries) if available from the electronic medical record. If SFDI correlates well with other clinical outcome assessments, it may be used in the future as a rapid, non-invasive tool for monitoring disease activity in scleroderma patients.

DETAILED DESCRIPTION:
The overall objective of this study is to determine if a light emitting diode (LED) -based SFDI instrument can be used to detect changes in skin thickness over time in SSc patients.

Number of subjects:

60 patients with scleroderma and 32 control subjects without scleroderma

Study procedures:

All subjects will have 6 areas of the body, right and left fingers, hands, and forearms, measured with an LED-based SFDI instrument every 3 months for the first 12 months and then every 6 months through 36 months. The right and left upper arms of subjects may be measured with the SFDI instrument if subjects are able to comfortably extend their arms.

All subjects will have the option to have blood collected for serum at baseline, 12 months, 24 months, and 36 months to investigate serum biomarkers of fibrosis.

An optional skin biopsy will be collected from all subjects at baseline, 12 months, 24 months, and 36 months to evaluate histopathological skin changes. Skin biopsies will not be collected from pregnant or lactating subjects, from subjects with a history of an allergic reaction to a local anesthetic, or from subjects who are deemed by the study doctor to be at high risk of small tissue calcification.

Scleroderma subjects will be asked to complete the SSPRO questionnaire at baseline and every 3 months for the first 12 months and then every 6 months through 36 months.

Scleroderma subjects will have a mRSS performed at baseline and every 3 months for the first 12 months and then every 6 months through 36 months.

All subjects will have durometry and ultrasound performed on the right and left forearms at baseline and every 3 months for the first 12 months and then every 6 months through 36 months.

Secondary Objectives:

* Assess how SFDI measurements correlate with other clinical measurements of skin thickness such as durometry, ultrasound, and mRSS
* Assess how SFDI measurements correlate with clinical biochemical and histopathological assessments of skin changes in SSc.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet at least one of the following:

* Have SSc as defined by the American College of Rheumatology (SSc subjects only)
* Suspected of having SSc based on clinical symptoms as determined by their physician (SSc subjects only)
* Defined as a healthy control (does not have SSc or another known disease that in the opinion of the investigator could confound the results)

Exclusion Criteria:

* Diagnosis of skin malignancy within the previous 2 years, excluding adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ.
* Presence of wounds or skin rashes at the site of Spatial frequency domain imaging (SFDI) measurement or skin biopsy
* Presence of other co-morbid illnesses with an estimated median life expectancy < 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Baseline SFDI measurements of skin thickness | baseline
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
6 months SFDI measurements of skin thickness | 6 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
12 months SFDI measurements of skin thickness | 12 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
18 months SFDI measurements of skin thickness | 18 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
24 months SFDI measurements of skin thickness | 24 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
30 months SFDI measurements of skin thickness | 30 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms
36 months SFDI measurements of skin thickness | 36 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms

SECONDARY OUTCOMES:
Serum fibrosis biomarkers, Chemokines that promote fibrosis | baseline and every 12 months up to 36 months
  Assessed from serum
Serum fibrosis biomarkers, Pro-inflammatory cytokines involved in immune cell migration | baseline and every 12 months up to 36 months
  Assessed from serum
Serum fibrosis biomarkers, Matricellular proteins | baseline and every 12 months up to 36 months
  Assessed from serum
histopathological assessments of skin collagen content | baseline and every 12 months up to 36 months
  Assessed from skin biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Bujor, MD, PhD, Principal Investigator — BU Chobanian & Advesian School of Medicine
Locations (1):
- Shapiro Outpatient Rheumatology Clinic at Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No